CLINICAL TRIAL: NCT06513325
Title: Association of Perceived Occupational Performance and Satisfaction, Balance, Gait, and Fear of Falling in Older Adult With Mild Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Güllü Aydın Yağcıoğlu, Assistant Professor, Gulhane School of Medicine
Other Study IDs: MCC-Geriatrics
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment; Gait; Balance; Occupational Problems
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Canadian Occupational Performance Measure — It is a semi-structured scale that helps to identify problematic areas of performance experienced by individuals and to measure their perceived occupational performance and satisfaction. This scale assesses the level of performance of self-care, productivity and leisureoccupations and satisfaction with these performances as perceived by the individual.

SUMMARY:
This study was designed to investigate the occupational performance and balance, gait, and fear of falling in older adults with MCI. Balance and gait of the older adults were assessed with the Tinetti balance and gait test, fear of falling with the Tampa Scale for Kinesiophobia and occupational performance with the Canadian Occupational Performance Measure (COPM). The relationship between COPM and other parameters was analysed by Spearmen's test.

ELIGIBILITY:
Inclusion Criteria:

* people over 65 with mild cognitive impairment who could understand and follow instructions

Exclusion Criteria:

* Individuals who were unable to participate in the study due to a chronic condition or the use of assistive devices such as wheelchairs or crutches

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study included people over 65 with mild cognitive impairment
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | 10 minutes
  It is a semi-structured scale that helps to identify problematic areas of performance experienced by individuals and to measure their perceived occupational performance and satisfaction. This scale assesses the level of performance of self-care, productivity and leisureoccupations and satisfaction with these performances as perceived by the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Güllü AYDIN YAĞCIOĞLU, Asst. prof, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aydin-Yagcioglu G, Ersoy K, Arslaner SB, Torpil B. Association between perceived occupational performance and satisfaction and balance, gait, and fear of falling in older adults with mild cognitive impairment. Br J Occup Ther. 2025 Jun 29;88(9):581-586. doi: 10.1177/03080226251340858. eCollection 2025 Sep. PMID 40893702